CLINICAL TRIAL: NCT06109636
Title: Correlation Analysis Between In-vivo Corneal Biomechanical Properties and Anterior Segment in Chinese Population
Brief Title: Correlation Analysis Between Corneal Biomechanics and Anterior Segment
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023025
Record Dates: First submitted 2023-10-21; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Ciliary Muscle Thickness; Anterior Sclera Thickness; Corneal Biomechanics; CASIA2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal group
  Interventions: Other: Pentacam, Corvis ST and Casia2

INTERVENTIONS:
Other: Pentacam, Corvis ST and Casia2 — scleral and ciliary muscle thickness were obtained by Casia2, biomechanical parameters were obtained by Pentacam and Corvis ST

SUMMARY:
Evaluation of the ciliary muscle thickness, area, and anterior chamber angle, as well as anterior sclera thickness in subjects, to investigate the relationship between these measurements and corneal biomechanics. Clarify whether aqueous humor displacement, anterior sclera, and ciliary muscles influence the assessment of in vivo corneal biomechanics.

ELIGIBILITY:
Inclusion Criteria:

1. Best corrected visual acuity (BCVA) ≥ 20/20;
2. No other eye diseases except myopia and astigmatism;
3. The cornea was transparent, and there was no cloud or pannus;

Exclusion Criteria:

1. Corneal disease;
2. Ocular trauma;
3. Previous ocular surgery;
4. Any anterior segment diseases except cataract;
5. Patients were required to stop wearing soft contact lenses for at least 2 weeks and rigid contact lenses for at least 4 weeks before examination;
6. Pregnant and lactating women;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients premedicated for refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-03-04 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
scleral and ciliary muscle thickness | one year
  The thickness of scleral and ciliary muscle(Casia2, quantitative data through the utilization of its integrated ruler system)
biomechanical parameters | one year
  The biomechanical parameters(Corvis ST, exporting the quality-assured csv files to analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Prof, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided